CLINICAL TRIAL: NCT01211938
Title: Randomized Phase 2 Trial Evaluating the Acute Toxicity of Two Protocols of Reirradiation After Surgery in an Irradiated Area for Carcinoma of the Upper Aerodigestive Tract - Single-fraction Radiotherapy With Concomitant 5FU and Hydrea Administered Every Other Week - Continuous Hyperfractionated Radiotherapy With Concomitant Cetuximab
Brief Title: Trial Comparing Two Protocols of re Irradiation in an Irradiated Area for Carcinoma of the Upper Aerodigestive Tract
Acronym: JANORL2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSET 1542-JANORL2; 2009-017047-34 (EudraCT Number)
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Squamous Cell Carcinoma
Keywords: phase II/III; upper aerodigestive tract carcinoma; re irradiation; Recurrent or second upper aerodigestive tract carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Recurrence | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single-fraction radiotherapy with concomitant 5FU and Hydrea (Active Comparator): six 5-day cycles with a 9-day rest period between each cycle (split course). Each cycle includes : a single-fraction at a dose of 2 Gy per session for 5 sessions, combined with 5FU (800 mg/m2/day) and Hydrea (500 mg x 3/day) over the 5 days of the cycle. The total dose of radiotherapy is therefore 60 Gy delivered over 11 weeks.
  Interventions: Radiation: single-fraction radiotherapy with concomitant 5FU and Hydrea
- hyperfractionated radiotherapy with concomitant Cetuximab (Experimental): Bifractionated radiotherapy at a dose of 1.2 Gy per session at a rate of 2 sessions per day, at least 6h apart, 5 days per week over 5 weeks, without a split course, combined with Cetuximab. The total dose of radiotherapy is 60 Gy delivered over 5 weeks. Cetuximab (ErbituxÒ) is to be administered in a 2-hour IV infusion at a dose of 400 mg/m2, 8 days before the start of radiotherapy, then in a 1-hour infusion at a dose of 250 mg/m2 on days 1, 8, 15, 22 and 29 of radiotherapy.
  Interventions: Radiation: hyperfractionated radiotherapy with concomitant Cetuximab

INTERVENTIONS:
Radiation: single-fraction radiotherapy with concomitant 5FU and Hydrea — single-fraction radiotherapy with concomitant 5FU and Hydrea
  Arms: single-fraction radiotherapy with concomitant 5FU and Hydrea
Radiation: hyperfractionated radiotherapy with concomitant Cetuximab — hyperfractionated radiotherapy with concomitant Cetuximab
  Arms: hyperfractionated radiotherapy with concomitant Cetuximab

SUMMARY:
Patients will be randomised after surgery, provided surgery is macroscopically adequate, that there is a flap of tissue protecting the vascular axis and that wound healing allows reirradiation to begin less than 8 weeks after surgery.Reirradiation will begin in the two arms less than 8 weeks after surgery in the irradiated area. The reirradiated volume : tumour bed + a safety margin of < 2 cm with immediate protection of bone marrow. This volume should be jointly defined by the radiotherapist and the surgeon. During reirradiation, 60 Gy will be delivered in the two arms but will last 11 weeks in the reference arm and 5 weeks in the investigational arm.Acute toxicity (NCI-CTCAE) will be evaluated at the end of reirradiation and at 6 months from randomization (first follow-up consultation)

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or second upper aerodigestive tract carcinoma in an area previously irradiated at a dose of >= 50 Gy
* Squamous cell carcinoma
* No grade III or IV sequels linked to the first radiation therapy (excepted radiation sequels of salivary glands)
* Relapse or second carcinoma (clinically invasive and/or lymph node recurrence >= 3 cm and/or the association of a local and lymph node recurrence
* Oral cavity, pharynx, larynx (if rT4), cervical region (if >3cm)
* No distant metastases confirmed by chest CT scan, abdominal ultrasound (or CT scan) in case of abnormal liver function, and bone scintigraphy in case of local symptoms
* Surgery in the previously irradiated region allowing a macroscopically adequate resection
* Surgery and vascular protection with a myocutaneous or free flap
* Interval > = 6 months between the end of the first radiation treatment and surgery in the previously irradiated area
* Wound healing allowing reirradiation within an interval of 8 weeks after surgery in the previouly irradiated area.
* No participation in a clinical trial during the 30 days preceding inclusion
* Age between 18 et 70 years.
* Performance Status 0 or 1 according to WHO criteria.
* Hematological function : neutrophils * 2 x 106/l, platelets : * 100 x 106/l, hemoglobin : * 10 g/dl (or 6.2 mmol/l)
* Liver function : total bilirubin (normal) ; ASAT (SGOT) and ALAT (SGPT) * 2.5 * upper limit of normal (ULN) in each centre ; alkaline phosphatases * 5 * ULN. Patients whose ASAT or ALAT levels > 1.5 * ULN associated with alkaline phosphatases * 2.5 * ULN are not eligible for the trial
* Renal function : serum creatinine * 120 *mol/l (1.4 mg/dl) ; if creatinine level is > 120 *mol/l, creatinine clearance should be * 60 ml/min.
* Written consent of participants

Exclusion Criteria:

* Superficial recurrence not associated with a lymph node relapse, isolated lymph node recurrence measuring less than 3 cm
* Distant metastases
* Grade 3 or 4 sequels of first radiation therapy (excepted salivary gland sequels)
* Macroscopically inadequate surgery
* Delay in wound healing obliging reirradiation to be postponed beyond 8 weeks.
* > Grade 3 Toxicity induced by chemotherapy administered during a previous treatment
* Hypersensitivity to Erbitux
* Concomitant severe comorbidities (non exhaustive list)
* Unstable cardiac comorbidity in spite of treatment.
* Neurological or psychiatric history such as dementia, convulsions.
* Severe uncontrolled infection
* Obstructive bronchopneumopathy which required hospitalisation during the year preceding inclusion.
* Factors (psychological, familial, social or geographic) likely to hinder patient compliance with the study protocol and follow-up are considered exclusion criteria. These factors should be discussed with the patient before enrollment in the trial
* Women who are pregnant, breast-feeding or of birthgiving age without effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2017-02-25 (Actual); Study Completion 2017-02-25 (Actual)

PRIMARY OUTCOMES:
Acute toxicity requiring an interruption of radiotherapy for more than 2 weeks | 6 months
Overall survival at 3 years and loco-regional control at 3 years | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- See also: ORL clinical trials on line in Institut Gustave Roussy — http://www.gustaveroussy.fr/fr/essai/cancers-orl-cancer-6